CLINICAL TRIAL: NCT03423394
Title: Improving Voluntary Engagement for PTSD Treatment Among Service Members
Brief Title: Efficacy Trial of Stress Check-Up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Denise Walker, Research Professor, School of Social Work, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00002794; W81XWH-17-1-0002 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2018-01-09; First posted 2018-02-06 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2021-09

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Motivational enhancement therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Motivational Interviewing; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Enhancement Therapy (Experimental): The MET intervention will consist of three 45-90 minute telephone delivered sessions that will be staggered to occur 1 week, 1 month, and 2 months after the baseline assessment.
  Interventions: Behavioral: Motivational Enhancement Therapy
- Treatment as Usual (Active Comparator): The treatment as usual (TAU) condition was selected to mirror the existing process in the military for identifying and encouraging treatment for personnel who screen positive for PTSD.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Motivational Enhancement Therapy — The MET intervention will consist of three 45-90 minute telephone delivered sessions that will be staggered to occur 1 week, 1 month, and 2 months after the baseline assessment. The first MET session intervention will involve a counselor using motivational interviewing (MI) strategies to establish an empathic therapeutic relationship and focus learning about the PTSD symptoms the participant is experiencing and exploring ambivalence about seeking treatment services. MET sessions 2 and 3 will focus on identifying and responding to risk factors for dropping out of treatment (increases in ambivalence, avoidance behavior, concerns about stigma, life chaos), identifying and responding to barriers to participant's active engagement in treatment, and facilitating enrollment in alternate therapeutic resources if necessary.
  Arms: Motivational Enhancement Therapy
Behavioral: Treatment as Usual — TAU will include a written referral list comprised of PTSD resources including information on in-person treatments, self-help, web-based and bibliotherapy options. At the completion of the study, participants in the TAU condition will be offered the MET intervention.
  Arms: Treatment as Usual

SUMMARY:
Untreated posttraumatic stress disorder (PTSD) is associated with high societal and individual costs. Effective interventions for symptoms of posttraumatic stress (PTS) exist but are underutilized by those who could benefit, especially among active duty military. This study will develop and test a brief telephone-delivered motivational enhancement intervention (MET) for military personnel (active, reserve, or national guard) serving in the Army, Air Force, or Navy who are experiencing symptoms of PTS, but who are not currently engaged in PTS treatment. The goal of the intervention is to decrease stigma around seeking care, increase knowledge about treatment options, increase engagement in help-seeking behavior, all leading to reductions in PTS symptoms.

DETAILED DESCRIPTION:
The health and well being of military personnel, and consequently the capacity for optimal functioning of military units, are compromised by posttraumatic stress disorder (PTSD). PTSD is associated with high personal and societal costs. Post-deployment rates of PTSD range from 5-20%; approximately 8% of combat exposed military personnel develop new onsets of PTSD. PTSD is frequently comorbid with other psychiatric disorders. Untreated PTSD is associated with high rates of suicide, medical services utilization, relationship impairment, legal difficulties, decreased worker productivity, and decreased military readiness.

While PTSD treatment can be effective, individuals with PTSD may not seek treatment. Drop out and medication noncompliance are common. Moreover, military personnel encounter both real and perceived barriers to seeking treatment. Given the availability of effective treatments contrasted with the low rates of military personnel who present and complete treatment, figuring out how to connect individuals with PTSD symptoms into treatment and then helping them to stay engaged is a high priority. Motivational enhancement therapy (MET) has shown promise in promoting treatment entry and enhancing both retention and successful outcomes. A brief, telephone-delivered MET called a "check-up," has shown promise in promoting self-initiated behavior change as well as voluntary treatment entry, enhanced retention, and more successful outcomes for substance abuse. Despite these promising findings, no work has focused on adapting MET for enhancing self-referral and treatment seeking with individuals with PTSD who are active duty and who are not already in treatment. Active duty military face additional challenges to entering treatment than veterans and thus specific research is necessary to evaluate whether similar programs would be efficacious for active duty personnel.

Adapting the "check-up" application with military personnel is warranted for three key reasons: (1) it has the potential of overcoming barriers to treatment-seeking, i.e., stigma and apprehension of a negative impact on one's military career; (2) it has the potential of attracting voluntary participation; and (3) protocols for disseminating this low cost intervention for use with deployed military can readily be developed and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Current PTSD
* Currently serving in the Army, Navy, or Air Force

Exclusion Criteria:

* Currently being treated (counseling and/or medication) for PTSD
* Non-fluency in English
* Evidence of psychosis
* Pending deployment that would preclude completion of follow-ups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) | 1 months
  The Clinician Administered PTSD Scale (CAPS) is a structured, clinician-administered interview that assesses the severity of each of the PTSD symptoms listed in Diagnostic and Statistical Manual of Mental Disorders (DSM-5) and yields a clinical PTSD diagnosis and overall severity rating. The CAPS total severity rating ranges from 0-80, with higher scores indicating greater PTSD severity.
Treatment Utilization | 3 months
  The Treatment Utilization questionnaire asks about current and past use of different treatment services.
  Part 1: Participants are asked (yes/no) if they have ever participated in treatment or support for different concerns (i.e., depression, marital or family concerns, posttraumatic stress, smoking cessation, anger management, and drinking or drug use) and then asked to identify type of treatment or support (i.e., self help, group therapy, individual therapy, medication, inpatient/ residential program, and other) they received for any of the concerns they reported "yes".
  Part 2: Participants are asked (yes/no/not applicable) if they have participated in treatment or support for any of the concerns reported in Part 1 in the past 3 months.
  Part 3: Participants are asked (yes/no) about their use of treatment and support resources used in the past 3 months for dealing with psychological or emotional concerns related to a traumatic event.
Treatment Reactions Scale | 3 months
  The Treatment Reactions Scale (TRS) is a 31-item measure that assesses the respondent's perceptions of treatment for mental and behavioral health. The TRS total score ranges from 31-155, with lower scores indicating more favorable reactions to treatment.
  The TRS consists of 5 subscales:
  Embarrassment/shame for seeking treatment (5 items, range 5-25; lower score indicates less embarrassment/shame for seeking treatment) Occupational/career impact of seeking treatment (4 items, range 4-20; lower score indicates less occupational/career impact of seeking treatment) Perceived debasement for receiving treatment (9 items, range 9-45; lower score indicates less perceived debasement for receiving treatment) Willingness to recommend treatment (7 items, range 7-35; lower score indicates more willingness to recommend treatment) Confidence in/belief in the efficacy of treatment (6 items, range 6-30; lower score indicates more confidence in/belief in the efficacy of treatment)

SECONDARY OUTCOMES:
Depression Module from the Patient Health Questionnaire (PHQ-9) | 2 weeks
  Measure that asks respondents to rate frequency of nine depressive symptoms over the past two weeks.
Daily Drinking Questionnaire | 1 week
  Measure that asks the respondent to think about a typical week and estimate the typical number of drinks he or she consumes each day of that week.
Alcohol Use Disorder Identification Test (AUDIT) | 6 months
  Measure that asks about the respondent's alcohol use.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington Innovative Programs Research Group, Seattle, Washington, United States

REFERENCES:
- [Derived] Walker DD, Walton TO, Jaffe AE, Graupensperger S, Rhew IC, Kaysen D. Improving voluntary engagement for posttraumatic stress disorder treatment among active-duty service members using motivational enhancement therapy. Psychol Trauma. 2024 Dec;16(Suppl 3):S492-S501. doi: 10.1037/tra0001562. Epub 2023 Oct 12. PMID 37824257
- [Derived] Jaffe AE, Walton TO, Walker DD, Kaysen DL. Social support and treatment utilization for posttraumatic stress disorder: Examining reciprocal relations among active duty service members. J Trauma Stress. 2023 Jun;36(3):537-548. doi: 10.1002/jts.22908. Epub 2023 Feb 2. PMID 36728194
- [Derived] Kaysen D, Walton TO, Rhew IC, Jaffe AE, Pierce AR, Walker DD. Development of StressCheck: A telehealth motivational enhancement therapy to improve voluntary engagement for PTSD treatment among active-duty service members. Contemp Clin Trials. 2022 Aug;119:106841. doi: 10.1016/j.cct.2022.106841. Epub 2022 Jun 28. PMID 35777697

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT03423394/Prot_SAP_000.pdf